CLINICAL TRIAL: NCT03506997
Title: PERSEUS1: Phase II Trial of the Immune Checkpoint Inhibitor Pembrolizumab for Patients Suffering From Metastatic Prostate Cancer
Brief Title: Trial of Pembrolizumab in Metastatic Castration Resistant Prostate Cancer
Acronym: PERSEUS1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICR-CTSU/2016/10060; 2017-000931-15 (EudraCT Number)
Record Dates: First submitted 2018-03-12; First posted 2018-04-24 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Castration-resistant Prostate Cancer
Keywords: Immune checkpoint inhibitor; Pembrolizumab
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Two stage Simon Minimax design phase II trial, with 90% power and 5% type I error to discard treatment if <20% responses are observed and detect activity >40%
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab will be given at a dose of 200mg IV every 3 weeks for a maximum of two years
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200mg given as a 30 minute intravenous (IV) infusion, on day 1 of each 3 week cycle. Patients may continue with pembrolizumab treatment as long as they remain free from intolerable toxicity for a maximum of two years, if in the Investigator's opinion they are receiving clinical benefit, and/or they do not meet any discontinuation criteria.
  Other Names: Keytruda; MK-3475

SUMMARY:
PERSEUS1 is an open-label, single arm, phase II trial evaluating the efficacy of Pembrolizumab in metastatic castration resistant prostate cancer (mCRPC) patients (Part A) with a biomarker enrichment stage (Part B) if efficacy is shown in part A.

DETAILED DESCRIPTION:
Open-label, single arm, phase II trial initially pursuing a two-stage Simon Minimax design. The null hypothesis Po will be 0.20; the alternative hypothesis Pa will be 0.40 (type 1 error will be 0.05 and type 2 error will be 0.10).

Patients with metastatic CRPC tumours characterised by high mutational load, high microsatellite instability as established, for example, by the Promega MSI 1.2 analysis system, or a DNA repair defect including loss of MMR, identified on archival or fresh tissue biopsy specimens (through a TMG approved sequencing study e.g. the MAESTRO study) who have either exhausted established active anticancer drugs, or preferred not to have established agents, will be offered entry into the PERSEUS1 study.

Part A: Part A is an open-label, single arm, two-stage Simon Minimax design phase II trial.

Stage 1: Patients will continue their LHRH analogue therapy. This cohort will include 24 patients as the first stage of a two-stage Phase II. If more than 5 responses in these first 24 patients are reported then the study will proceed to stage 2. Anti-tumour activity will be assessed (measured by response rates) by PSA, imaging assessments (CT & bone scans or when indicated whole body MRI) and CTC count measures. Whole Body MRI (WB-MRI) will be performed instead of CT in patients with contraindications to CT contrast), or instead of bone scan in patients with widespread bone disease at baseline thought to be non-evaluable by PCWG criteria due to inability to reliably identify two new lesions.

Stage 2: This will enrol a further 21 patients to a total of 45 patients. Ineffectiveness will be concluded if ≤5 and ≤13 responses are seen in the stage 1 and stage 2 respectively and the null hypothesis will be rejected (i.e. further research would be warranted) if >13 responses are reported from the first 45 patients.

With this Simon Minimax design the probability of early termination of this trial when the true response probability (P0) is <0.20 is 0.66.

Part B: Biomarker enrichment stage: If the null hypothesis is rejected (and with Sponsor approval and confirmation of sufficient funding) the study will continue with stratified recruitment into biomarker defined cohorts in order to increase the precision with which the response rate can be estimated within mCRPC molecular subgroups of interest. It is anticipated that approximately 55 patients will be included in Part B, which will make a total of 100 mCRPC patients in part A and B together, including ≥9 patients for each of:

A) MMR defective mCRPC; B) High mutational load mCRPC without MMR defects; C) mCRPC with deleterious homologous recombination (HR) DNA repair aberrations (BRCA2, ATM, BRCA1, PALB2, others); D) mCRPC with deleterious nucleotide excision repair (NER) aberrations; E) mCRPC with deleterious base excision repair (BER) aberrations; F) mCRPC with deleterious aberrations in non-homologous end-joining (NHEJ).

Eligibility for more than one cohort is anticipated to be uncommon; where this occurs "allocation" to a cohort will be determined in discussion with the CI based on initial sequencing results and with priority given to driver (rather than sub-clonal) mutations. Patients recruited in Part A will be retrospectively "allocated" to a cohort on the basis of their initial sequencing data (reported prior to trial entry) prior to any response assessments, for the purposes of analysis. Within each biomarker subgroup (A-F) this will allow us to reject the probability of a >30% response rate if we see no responses in 9-patients, with a 5% false negative risk (Gehan design). If ≥1 responses are seen in 9 patients in a subtype, recruitment will continue to that subtype with a further 20-25 patients such that the final estimate of the response rate has a standard error of 10%. Response rates with confidence intervals will be reported for each subtype.

In the absence of any safety concerns from the IDMC, recruitment will continue seamlessly from Part A stage 1 to Part A stage 2 and from Part A stage 2 to the Part B biomarker enrichment cohorts. It is possible that at the time of the Part A stage 1 and 2 overall analysis (based on 45 patients), the graduation of some of the more common subgroups to the enrichment phase will be known (e.g. if more than 1 response from 9 patients recruited to a biomarker subgroup that cohort would continue to at least 20 patients). Conversely, if no successes have been seen in 9 patients of a particular subtype, recruitment to that subtype would not proceed to the enrichment stage.

The biomarker defined cohorts may accrue at different rates related to genomic prevalence. At each stop/go decision point (end of enrichment stage 1 in a particular cohort) overall progress of all the ongoing enrichment cohorts will be reviewed by the IDMC/TSC. They will be asked to advise on the value of continued accrual to the cohorts particularly in light of slow recruitment.

ELIGIBILITY:
Inclusion Criteria:

1. Male, aged 18 years or older.
2. Histologically confirmed metastatic castrate resistant adenocarcinoma of the prostate. If the patient does not have a prior histological diagnosis then the planned baseline fresh biopsy may be used for both the purpose of confirming the histological diagnosis prior to trial entry and for subsequent biomarker analysis. All patients must be willing to have fresh biopsies to obtain tumour tissue for biomarker analysis.
3. Identified high mutational load (defined as 11 or more mutations per targeted panel - see Section 5.5 below) on next generation sequencing and/or a DNA repair defect that can increase mutation load including MMR deficiency and/or high MSI by next generation sequencing.
4. Patients with no measurable disease and only widespread bone disease must have a CTC count >5.
5. Willing and able to comply with the follow-up schedule and the requirements of the biomarker studies including the paired fresh tumour biopsies.
6. Written informed consent.
7. Prior treatment with at least one of the approved treatments for mCRPC (i.e. Abiraterone, Enzalutamide, Docetaxel, Cabazitaxel, Radium 223).
8. At least 28-days washout at trial entry since the completion of prior therapy, including major surgery, chemotherapy and other investigational agents. For hormonal treatment and radiotherapy refer to the guidelines below:

   • At least 28-days since the completion of prior flutamide treatment. Patients whose PSA did not decline in response to antiandrogens given as a second line or later intervention will only require a 14-day washout prior to Cycle 1, Day 1.
   * At least 42-days since the completion of prior bicalutamide (Casodex) and nilutamide (Nilandron) treatment. Patients whose PSA did not decline for at least 3-months in response to antiandrogens given as second line or later intervention will require only a 14-day washout period prior to Cycle 1 Day 1.
   * At least 14-days from any radiotherapy with the exception of a single fraction of radiotherapy for the purposes of palliation (confined to one field) is permitted.
9. Documented prostate cancer progression as assessed by the investigator with one of the following:

   • PSA progression defined by a minimum of three rising PSA levels with an interval of ≥ 1-week between each determination. The PSA value at the Screening visit should be ≥ 2 µg/L (2 ng/ml) if there is no measurable disease; patients on systemic glucocorticoids for control of symptoms must have documented PSA progression by PCWG3 while on the same dose of systemic glucocorticoids prior to commencing Cycle1 Day1 of treatment.

   • Radiographic progression of soft tissue disease by iRECIST criteria or of bone metastases by PCWG3 criteria with two or more confirmed new bone lesions on a bone scan/wb-MRI with or without PSA progression.
10. Surgically or medically castrated, with testosterone levels of <50 ng/dL (<2.0 nM). If the patient is being treated with LHRH agonists (patient who have not undergone orchiectomy), this therapy must have been initiated at least 4 weeks prior to Cycle 1 Day 1 and must be continued throughout the study.
11. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
12. Albumin ≥25 g/L.
13. Patient and the patient's partner of reproductive potential who are sexually active, must agree to use adequate methods of contraception during the course of the study and for 120 days after the last dose of study drug (see appendix A3 for accepted methods of contraception).
14. QT interval corrected for heart rate according to Fridericia's formula (QTcF) <470 msec or <480 msec with bundle branch block.
15. Patients with primary hypothyroidism can be considered eligible if thyroid stimulating hormone (TSH) at the screening visit is within normal range while patient is under hormonal treatment.
16. Subjects must have adequate bone marrow, hepatic and renal function documented within 7-days of trial entry defined as:

Haemoglobin (Hb) ≥ 9.0 g/dL Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L Platelet count ≥ 100 x 10^9/L International normalised ratio (INR) ≤ 1.5x upper limit of normal (ULN) Or: Prothrombin time ≤ 1.5x upper limit of normal (ULN) Serum bilirubin (for patients with total bilirubin >1.5x ULN) Or: Direct bilirubin ≤ 1.5x ULN ≤1.5x ULN Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5x ULN (for patients with liver metastases ≤ 5x ULN is permissible) Serum creatinine ≤1.5 x ULN Or: Calculated creatinine clearance >40mL/min for patients with creatinine levels above institutional normal. For GFR estimation, the Cockcroft and Gault equation should be used: creatinine clearance = (((140 - age) x mass (kg)) x 1.23) / serum creatinine (µ mol⁄L)

Exclusion Criteria:

* 1. Patients with a history of prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-OX-40, anti-CD40, or anti-CTLA-4 antibodies.

  2. Patients who have received any of the following concomitant therapies: IL-2, interferon or other non-study immunotherapy regimens; immunosuppressive agents; other investigational therapies; or chronic use of systemic corticosteroids (used in the management of cancer or non-cancer-related illnesses) within 1 week prior to first dose. A dose of 10mg of prednisolone or equivalent will be allowed if clinically indicated.

  3. Patients who have received any non-oncology vaccine therapy used for prevention of infectious diseases including seasonal vaccinations for up to 28-days prior to the expected start or after any dose of pembrolizumab. Examples include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, seasonal flu, H1N1 flu, rabies, BCG, and typhoid vaccine.

  4. Patients receiving growth factors including, but not limited to, granulocyte colony stimulating factor (G-CSF), granulocyte macrophage-colony stimulating factor (GM-CSF), erythropoietin, within 14-days of study drug administration. Use of such agents while on study is also prohibited. Prior use of growth factors should be documented in the patient's medical history.

  5. Uncontrolled intercurrent cardiovascular disease as symptomatic congestive heart failure (New York Heart Association Class III or IV heart disease), unstable angina pectoris, cardiac arrhythmia, poorly controlled hypertension (defined as systolic blood pressure of ≥150mmHg or diastolic blood pressure of >100 mmHg based on a mean of three measurements at approximately 2-minute intervals).

  6. Any psychiatric illness/social situations that would limit compliance with study requirements.

  7. Any acute toxicity due to prior chemotherapy and / or radiotherapy that has not resolved to a NCI-CTCAE v4 grade ≤1 with the exception of chemotherapy induced alopecia and grade 2 peripheral neuropathy.

  8. Prior malignancy diagnosed within the previous 2-years with a >30% probability of recurrence within 12-months, with the exception of non-melanoma skin cancer, and in-situ or non-muscle invasive bladder cancer.

  9. Patients with myelodysplastic syndrome or acute myeloid leukaemia. 10. Patients with known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.

  11. Patients with symptomatic or impending cord compression unless appropriately treated beforehand and clinically stable and asymptomatic.

  12. Any chronic respiratory disease. 13. Any immunological disorder requiring treatment with immunosuppressive treatments:

  • High dose of steroids (low dose of steroids as 10mg of prednisolone or equivalent are allowed if the patient is not able to discontinue this treatment; patient needs to be on a stable dose for at least 4-weeks before the enrolment);
  * Cytotoxic agents (such as alkylating agents or antimetabolites);
  * Antibodies (polyclonal antibodies; monoclonal antibodies different from pembrolizumab);
  * Drugs acting on immunophilins (cyclosporin, tacrolimus, sirolimus);
  * Other drugs (interferons, TNF binding proteins, mycophenolate). 14. History of any autoimmune disease: patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]); CNS or motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre syndrome and myasthenia gravis, multiple sclerosis). Patients with controlled Graves' disease will be allowed.

    15. Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies). 16. Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).

    17. History of congenital platelet function defect (e.g., Bernard-Soulier syndrome, Chediak-Higashi syndrome, Glanzmann thrombasthenia, storage pool defect).

    18. Patients with history of (non-infectious) pneumonitis that required steroids or current pneumonitis.

    19. Initiating bisphosphonate therapy or adjusting bisphosphonate dose/regimen within 30 days prior to Cycle 1 Day 1. Patients on a stable bisphosphonate regimen are eligible and may continue.

    20. Presence of a condition or situation, which, in the investigator's opinion, may put the patient at significant risk, may confound the study results, or may interfere significantly with the patient's participation in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-11-27 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate tumour response | 6 months post trial entry
  Responses will be defined on the basis of the following outcomes; if any of these occur patients will be considered to have responded:
  * Objective response by iRECIST 1.1;or
  * CTC count conversion from >5 to <5
  * PSA decline of ≥50%. Responses will need confirmation by a second consecutive value obtained four or more weeks after the first value indicated a response. Evaluable patients with no confirmed response as defined above will be classified as non-responders. Response will be evaluated 6 months post-trial entry. The last value of PSA, CTC count, CT scan/bone scan/WB-MRI on or up to 28 days before the date of first study treatment will be used as the baseline value for this assessment.

SECONDARY OUTCOMES:
Radiological progression-free survival (rPFS) | From date of randomisation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  rPFS will be measured from the date of trial entry to the first occurrence of radiological progression or death from any cause. If no event exists then rPFS will be censored at the last scheduled disease assessment on study.
Time to radiological progression | From date of randomisation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Death from prostate cancer or any other cause without prior radiological evidence of progression will not count as an event. If no event exists, then time to radiological progression will be censored at the last scheduled disease assessment on study or date of disease whichever occurs earlier.
Progression free survival | From date of randomisation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  If no event exists, then PFS will be censored at the last scheduled disease assessment on study
Time to PSA progression | From date of randomisation until the date of first documented PSA progression or date of death from any cause, whichever came first, assessed up to 100 months
  PSA progression is defined according to the PCWG3 guidelines and is the date that a ≥ 25% increase and an absolute increase of ≥ 2 ng/mL above the nadir (baseline if no decline) is documented. This must be confirmed by a second consecutive value obtained 4 or more weeks later.
Duration of PSA response | From date of first decline by at least 50% until the time time there is an increase of 25% of PSA nadir or date of death from any cause, whichever came first, assessed up to 100 months
  calculated from the time the PSA value first declines by at least 50% of the cycle 1 day 1 (baseline) value (must be confirmed by a second value) until the time there is an increase of 25% of PSA nadir, provided the absolute increase is at least 2 ng/mL. The increase must be confirmed by a second consecutive measurement that is at least 25% above the nadir. If the PSA never shows a 25% increase over the nadir value, then the patient will be assessed at the last PSA measurement. PSA objective response rate (PSA-ORR) is calculated as the proportion of evaluable patients who achieve a PSA response.
Overall survival | From date of randomisation until the date of death from any cause, assessed up to 100 months
  Survival time of living patients will be censored on the last date a patient is known to be alive or lost to follow-up.
Safety and tolerability defined by CTC-AE, V 4.0 criteria. | From date of randomisation until the end of treatment or date of death from any cause, whichever came first, assessed up to 36 months
  Adverse events will be summarised by grade according to the worst grade experienced. In addition, the most frequently observed AEs will be summarised.

OTHER OUTCOMES:
Exploratory: • Molecular endpoints from both diagnostic archival FFPE tumour tissue (when available) and fresh mCRPC tumour tissue | From date of randomisation until the end of trial or date of death from any cause, whichever came first, assessed up to 100 months
  PD-1, PDL-1 and PDL-2 expression
Exploratory: • Molecular endpoints from both diagnostic archival FFPE tumour tissue (when available) and fresh mCRPC tumour tissue | From date of randomisation until the end of trial or date of death from any cause, whichever came first, assessed up to 100 months
  T-Reg infiltration (CD4+ CD25+ FoxP3+)
Exploratory: • Molecular endpoints from both diagnostic archival FFPE tumour tissue (when available) and fresh mCRPC tumour tissue | From date of randomisation until the end of trial or date of death from any cause, whichever came first, assessed up to 100 months
  CD3, CD8, lymphocyte infiltration
Exploratory: • Molecular endpoints from both diagnostic archival FFPE tumour tissue (when available) and fresh mCRPC tumour tissue | From date of randomisation until the end of trial or date of death from any cause, whichever came first, assessed up to 100 months
  Presence of mismatch repair defect as determined by immunohistochemistry or microsatellite instability (MSI).
Exploratory: • Molecular endpoints from both diagnostic archival FFPE tumour tissue (when available) and fresh mCRPC tumour tissue | From date of randomisation until the end of trial or date of death from any cause, whichever came first, assessed up to 100 months
  Mutational load (number of mutations per MB of DNA sequenced)
Exploratory: next generation sequencing data | From date of randomisation until the end of trial or date of death from any cause, whichever came first, assessed up to 100 months
  NGS data from tumour DNA and RNA including analyses of neoepitopes by targeted panel NGS and exome/transcriptome analyses when feasible.
Exploratory: Immunophenotyping endpoint | From date of randomisation until the end of trial or date of death from any cause, whichever came first, assessed up to 100 months
  WBC immunotyping
Exploratory:Whole blood mRNA expression profiling | From date of randomisation until the end of trial or date of death from any cause, whichever came first, assessed up to 100 months
  Whole blood mRNA expression profiling
Exploratory: Immune cell genomics including T-cell receptor sequencing | From date of randomisation until the end of trial or date of death from any cause, whichever came first, assessed up to 100 months
  Immune cell genomics including T-cell receptor sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Johann de Bono, Principal Investigator — The Institute of Cancer Research/The Royal Marsden NHSFT
Locations (1):
- The Royal Marsden Hospital, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided